CLINICAL TRIAL: NCT05309954
Title: Genetic Analysis to Predict the Development of Paget's Disease
Acronym: GAPDPD
Status: Active, not recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: European Research Council (Other)
Responsible Party: Sponsor
Other Study IDs: AC19056; 19/ES/0141 (Other: [Research Ethics Committee (EoSRES)); 259285 (Other: IRAS (Integrated Research Application System))
Record Dates: First submitted 2022-03-11; First posted 2022-04-04 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Paget Disease; Paget Disease of Bone
MeSH Terms: conditions — Osteitis Deformans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples, saliva samples and stool samples will be collected from participants in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational (With Bone Scan): Individuals with a Family history of Paget's disease of bone (PDB) affecting first degree relative such as a parent or sibling that have not already diagnosed with PDB
- Observational (Without Bone scan): Individuals, that are spouses, friends and/or non blood relatives of the individuals with a family history of PDB.

SUMMARY:
Paget's disease of the bone (PDB) is a skeletal disorder with a strong genetic component which can be associated with various complications such as pain, bone deformity, arthritis and deafness. Recent advances in understanding the genetic determinants of PDB offer the prospect of developing a genetic profiling test which can be offered to people with a parent or sibling with PDB to determine how likely they are to develop the disease themselves.

The aim of the study is to perform genetic testing for variants associated with PDB in people aged 45 and above who have a parent or sibling (first degree relative) with the disease. The Investigators will assess how well genetic profiling performs in predicting PDB by performing an imaging technique called a radionuclide bone scan which is a very sensitive way of detecting early PDB. This scan will be performed on entry to the study and again after five years. The reason for performing two scans five years apart because PDB becomes more common with age and so this will allow the Investigators to give an accurate indication of how good the genetic profiling test is in people at different ages. In addition to genetic profiling the investigators will analyse blood samples for biochemical markers of PDB and also test saliva and stool samples for the microbiome profile since its thought that this may influence risk of the disease as well.

In the longer term the investigators hope the study will allow them to develop a blood test to stratify for risk of PDB and use bone scans only in people who the clinicians think are at highest risk of developing the disease. This will allow people with PDB to be picked up early allowing treatment to be given in a timely manner.

DETAILED DESCRIPTION:
Paget's disease of bone (PDB) is a common skeletal disorder characterised by increased bone turnover affecting one or more bones throughout the skeleton. The natural history of PDB is incompletely understood but it is clear that patients are often asymptomatic when the disease is at an early stage but that later in life when the patient presents clinically, irreversible skeletal damage is often present leading to various complications, some of which are irreversible. The most common symptom of PDB is bone pain which can be due to increased metabolic activity or complications such as bone deformity, secondary osteoarthritis, spinal stenosis and pathological fractures. Other complications include deafness due to involvement of the temporal bone and osteosarcoma which is rare but often fatal.

Genetic factors play an important role in PDB and people who have a family history of the disease in a first- degree relative have a seven-times increased risk of developing the disease as compared with controls. Part of the genetic risk for developing PDB is explained by inheritance of mutations in the SQSTM1 gene. Cross-sectional studies indicate that carriers of SQSTM1 mutations run a high risk of developing the disease with increasing age. However only 40% of people with a family history of PDB carry SQSTM1 mutations and current evidence suggests that the risk of PDB in people who do not carry SQSTM1 mutations is mediated by inheritance of other susceptibility alleles which individually have modest effects on the risk of developing PDB but which when combined, have additive effect on disease susceptibility. Environmental factors also play a role in PDB and in keeping with this a recent study has shown that epigenetic factors contribute to the pathogenesis of PDB and may have value as diagnostic markers for the risk of developing the disease.

It would be highly advantageous to be able to offer people with a family history of PDB a predictive test to give an indication of their personal risk of PDB. This would allow the disease to be picked up at an early stage before complications have occurred and for preventative treatment to be offered. Prevention is key since there is no evidence that treatment can prevent or reverse complications in people with established disease.

The aim of the present study is to try and identify genetic, epigenetic and other biomarkers for the development of PDB in people with a family history of the disorder in order to facilitate early diagnosis and treatment.

ELIGIBILITY:
INCLUSION CRITERIA CASES

* Family history of PDB affecting first degree relative such as a parent or sibling.
* Not already diagnosed with PDB
* Participant willing and able to consent and comply with the study protocol.
* Age > 45 at the time of enrolment.

EXCLUSION CRITERIA CASES

* Unable or unwilling to provide informed consent
* Contraindication to radionuclide bone scan
* Already diagnosed with PDB

INCLUSION CRITERIA CONTROLS

* Spouse, partner or friend of case
* Not diagnosed with PDB
* No family history of PDB
* Participant willing and able to consent and comply with the study protocol.
* Age > 45 at the time of enrolment

EXCLUSION CRITERIA CONTROLS

• Unable or unwilling to give informed consent

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will aim to recruit up to individuals (Cases) with a positive family history of PDB and Spouses, friends and or unrelated relatives of the cases as a control cohort.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
PRIMARY ENDPOINTS - Identify Genetic Markers that are associated with the increased presence of PDB lesions in people with a family history of the disorder, as assessed by a radionuclide bone scan | 5 years
  Genetic and Transcriptome profile of each participant will be produced and analysed to determine if there is any association between specific genes and a increase in the presence of PDB lesions in people with a family history of the disorder. PDB lesions will be assessed by a radionuclide bone scan
Primary Endpoint (Participant arm): The proportion of patients that develop PDB-like bone lesions | 5 years
  The proportion of participants who have a family history of PDB that develop PDB-like bone lesions by the end of study assessed by radionuclide bone scan.
Primary Endpoint (Participant arm): T proportion of individuals that develop abnormalities suggestive of PDB | 5 years
  The primary endpoint will be to evaluate the proportion of individuals that develop biochemical or clinical abnormalities suggestive of PDB over a the 5-year duration of the trial

SECONDARY OUTCOMES:
Secondary Endpoint - Analysis of scores in SF36 (36-Item Short Form Survey) | 5 years
  SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. Scoring is a two-step process. First, precoded numeric values are recoded per a scoring key. Note that all items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved. In step 2, items in the same scale are averaged together to create a scale of scores.
  Analyse the difference in scores between Participant and control groups with regard to SF36 (36-Item Short Form Survey) scores. Scores associated with Health-related quality of life, Depression, anxiety and pain will be analysed and compared between the two groups
Secondary Endpoint- Analysis of scores in HAQ (Health Assessment Questionnaire) | 5 years
  the HAQ assesses a patient's level of functional ability and includes questions of fine movements of the upper extremity, locomotor activities of the lower extremity, and activities that involve both upper and lower extremities. There are 20 questions in eight categories of functioning which represent a comprehensive set of functional activities. The participant's responses are made on a scale from zero (no disability) to three (completely disabled).
  Analyse the HAQ (Health Assessment Questionnaire) scores to determine if there is a differences between Participant and control groups. Scores associated with Health-related quality of life will be analysed and compared between the two groups
Secondary Endpoint - Analysis of scores in EQ5D (EuroQol five dimension scale) | 5 years
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. . Each level is rated on scale that describes the degree of problems in that area also has an overall health scale where the rater selects a number between 1-100 to describe the condition of their health, 100 being the best imaginable.
  Analyse the EQ5D (EuroQol five dimension scale) scores to determine if there is a differences between Participant and control groups. Scores associated with Health-related quality of life, Depression, anxiety and pain will be analysed and compared between the two groups
Secondary Endpoint - Analysis of scores in IPAQ (International Physical Activity Questionnaire) | 5 years
  The IPAQ form is an instrument designed primarily for population surveillance of physical activity among adults. IPAQ assesses physical activity undertaken across a comprehensive set of domains Continuous Score Expressed as MET-min per week: MET level x minutes of activity x events per week Sample Calculation MET levels MET-min/week for 30 min episodes, 5 times/week Walking = 3.3 METs 3.3*30*5 = 495 MET-min/week Moderate Intensity = 4.0 METs 4.0*30*5 = 600 MET-min/week Vigorous Intensity = 8.0 METs 8.0*30*5 = 1,200 MET-min/week ___________________________ TOTAL = 2,295 MET-min/week Total MET-min/week = (Walk METs*min*days) + (Mod METs*min*days) + Vig METs*min*days). A higher MET value would be indicative of more activity during that week.
  Analyse the IPAQ scores to determine if there is a differences between Participant and control groups.
Secondary Endpoint - Analysis of scores in BPI (Brief Pain Inventory Scale) scores. | 5 years
  The Brief Pain Inventory (BPI) is a self-administered assessment tool used in pain management. The BPI uses simple numeric rating scales (NRS) from 0 to 10, and the scale defines pain as follows: Score: 1 - 4 = Mild Pain, Score: 5 - 6 = Moderate Pain, Score: 7 - 10 = Severe Pain.
  Analyse the BPI (Brief Pain Inventory Scale) scores to determine if there is a differences between Participant and control groups.
Secondary Endpoint- Specialised Biomarker Analysis | 5 years
  Samples from both Participants and control group would be analysed for Specialised Biomarkers of Bone turnover (P1NP, BSALP, uNTx CTx). Activity of these markers will be analysed and compared between the two cohorts to determine if there is a difference and if it can be used a predictor

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Ralston, Principal Investigator — University of Edinburgh
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided